CLINICAL TRIAL: NCT06642259
Title: Correlation Between Triglyceride Glucose Index and Residual SYNTAX Score in ST-elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Correlation Between Triglyceride Glucose Index and Residual SYNTAX Score in STEMI Patients Undergoing PPCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohammad medhat elsayed hasan, Assistant Lecturer, Assiut University
Other Study IDs: (TyG) index and SYNTAX
Record Dates: First submitted 2024-09-18; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Echocardiography — ECHO

SUMMARY:
The goal of this study To check correlation between triglyceride glucose (TyG) index and residual SYNTAX score (RSS) in STEMI patients undergoing PPCI.

2. Impact of both TyG index and RSS in STEMI patients undergoing PPCI on LV EF recovery after 3 months using LV speckle tracking.

3. Impact of RSS and TyG index in STEMI patients undergoing PPCI on short term MACE at 3 months duration.

DETAILED DESCRIPTION:
ST-elevation myocardial infarction (STEMI) is known as a life-threatening complication of coronary artery disease (CAD) and it is one of the leading causes of death all over the world. Primary percutaneous coronary intervention (PPCI) of the culprit vessel in patients with STEMI is standard clinical practice .

At the time of PPCI, 40-65% of the patients exhibit one or more concomitant coronary lesions (i.e., multivessel disease (MVD)). The presence of narrowed coronaries other than those related to index ischemia in patients with STEMI is suggested as a feature associated with adverse clinical outcomes .

The recently developed residual SYNTAX Score (RSS) (developed 2012 and validated in 2013) is an objective, quantitative measure of the degree and complexity of residual stenosis after percutaneous coronary intervention (PCI) .It was developed to quantitatively assess the degree and complexity of residual stenoses, based on recalculating the SYNTAX score from coronary angiography after PCI . Higher RSS has been associated with worse outcome in patients undergoing angiography-mediated PCI .

Insulin resistance (IR) is an important risk factor for the development of CAD . It is defined as a state in which a greater than normal amount of insulin is required to elicit a quantitatively normal response .

Previous studies have shown an independent association between IR and CVD. IR is tightly associated with increased cardiovascular morbidity and mortality by adversely modifying well-established cardiovascular risk factors such as dyslipidemia and hypertension and by causing endothelial dysfunction .

ELIGIBILITY:
Inclusion Criteria:

* All patient who are between 18 and 80 years old who present to our hospital (Assiut university heart hospital) with STEMI and eligible for primary PCI as treatment of choice according to guidelines, will be included in our study.

Exclusion Criteria:

* Patient who refuse to undergo revasculariztion using primary PCI.
* Patient who will die before withdraw of laboratory blood sample.
* Patient with previous PCI and/or CABG.
* Patient with underlying co-morbidity with life expectancy less than 1 year (end stage liver disease, end stage renal disease on regular dialysis, active malignancy).
* Patient with failed canalization of infarct related artery.
* Patient referred to CABG after angiography.
* Patient who is unconscious after cardiac arrest .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with STEMI and will undergo PPCI and fulfilling our inclusion criteria over a period of 6 months will be enrolled in our study.
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
1. To check correlation between triglyceride glucose (TyG) index and residual SYNTAX score (RSS) in STEMI patients undergoing PPCI | baseline
  1. To check correlation between triglyceride glucose (TyG) index and residual SYNTAX score (RSS) in STEMI patients undergoing PPCI.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Roshdy, Pro, Study Director — Assiut University